CLINICAL TRIAL: NCT01018056
Title: Developing New Treatments for Tourette Syndrome: Therapeutic Trials With Modulators of Glutamatergic Neurotransmission
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00023969; R34MH085844 (NIH)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; glutamatergic therapy; D-serine; riluzole; glutamate; glutamate agonist; glutamate antagonist; Tourette syndrome treatment study; OCD; tics
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- D-serine (glutamate agonist) (Experimental): 24 subjects age 8-17 years with moderate to severe TS (TTS > 22) will be enrolled in this treatment arm. They will receive D-serine for 6-weeks of the study, during which time drug dose may gradually be increased as needed. At 6-weeks participants will taper off drug.
  Interventions: Drug: D-serine
- Riluzole (glutamate antagonist) (Experimental): 24 subjects age 8-17 years with moderate to severe TS (TTS > 22) will be enrolled in this treatment arm. They will receive riluzole for 6-weeks of the study, during which time drug dose may gradually be increased as needed. At 6-weeks participants will taper off drug.
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator): 12 subjects age 8-17 years with moderate to severe TS (TTS > 22) will be enrolled in this treatment arm. They will receive placebo for 6-weeks of the study, during which time drug dose may gradually be increased as needed. At 6-weeks participants will taper off drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-serine — The dosage schedule will be flexible with a maximum dose for each subject being 30 mg/kg/day. In any individual subject, dose escalation may proceed more slowly, or the dose may be reduced if necessary. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of capsules labeled as study drug, but containing either 250 or 500 mg tablets of D-serine or placebo; capsule content to be determined by patient's weight. No changes in dosage will be made during the final week of treatment.
  Arms: D-serine (glutamate agonist)
Drug: Riluzole — The starting dose of riluzole will be 50 mg for one week; administered as one capsule (50) every morning. Dosage schedules will be flexible. If needed for tic suppression, the dose will be increased weekly by 50 mg and given in BID doses. The maximum dose will be 200 mg/day (administered as 2 capsules BID). In any individual subject, dose escalation may proceed more slowly, or the dose may be reduced if necessary. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing placebo capsules. No changes in dosage will be made during the final week of treatment.
  Other Names: Rilutek
  Arms: Riluzole (glutamate antagonist)
Drug: Placebo — Placebo tablets will be formulated in look-alike capsules. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing additional placebo capsules.
  Arms: Placebo

SUMMARY:
A joint NIH -Tourette Syndrome Association Conference has emphasized the critical need for the testing and development of new pharmacotherapy for tic suppression in Tourette syndrome (TS). This submission is a safety, tolerability and efficacy pilot study using two medications that modulate glutamate neurotransmission, riluzole, a glutamate antagonist, and D-serine, a glutamate agonist. Glutamate is the primary excitatory neurotransmitter in the central nervous system, an essential component of pathways implicated in TS and an extensive modulator of dopamine, the major neurotransmitter associated with tics.

This is a single site, short-term, proof of concept study of riluzole and D-serine for the treatment of tics. Each medication will be evaluated and compared to placebo as part of a double-blind, randomized, parallel, flexible dose, three-arm, 8-week, treatment protocol (D-serine, riluzole, or placebo). A total of sixty patients (age 8-17 years) with TS and moderate to moderately-severe tics will receive study medication according to a 2:1 (dopamine modulating drug: placebo), randomized schedule, i.e., riluzole (n=24), D-serine (n=24), placebo (n=12). The primary outcome measure is tic suppression as determined by changes in the Total Tic Subscore of the Yale Global Tic Severity Scale (YGTSS). Secondary tic outcome measures include changes in the YGTSS Total Score and two Global Impression Scales. Further, since both riluzole and D-serine have been proposed as treatments for obsessive-compulsive behaviors, a TS co-morbidity, these symptoms will be followed. Safety measures include serial physical examinations, vital signs, laboratory studies (comprehensive metabolic panel, complete blood count, plasma amino acids, and urine analyses), documentation of side effects and adverse events, and measurement of changes in ADHD, depression and anxiety.

This pilot investigation will provide important proof-of-concept data on glutamate therapies for TS and, in turn, evidence for large-scale, multi-center clinical trials.

DETAILED DESCRIPTION:
Study Design Overview: The goal of this study is to perform a short-term, proof of concept study to examine the safety, tolerability and efficacy of riluzole and D-serine in the treatment of tics. Each medication will be evaluated and compared to placebo as part of a randomized, double-blind, flexible dose, parallel, eight-week protocol, containing six weeks of active treatment (D-serine, riluzole, or placebo). A total of sixty patients (age 8-17 years) with Tourette syndrome or chronic motor tics (Tourette Syndrome Study Group criteria) having moderate to moderately-severe tics will participate; riluzole (n=24), D-serine (n=24), placebo (n=12).

This study contains six weeks of active treatment with D-serine, riluzole or placebo. The decision to implement a 6-week treatment protocol was based on the following: a) the ability to gradual increase doses of medication on a weekly basis over the first five weeks to dosages beneficial in other conditions; b) a treatment duration similar to that used in other glutamate modulatory treatment studies; and c) a time period necessary to identify a treatment effect in milder non-neuroleptic tic-suppressing medications such as clonidine. We emphasize that this is a short term, proof of concept study for riluzole and D-serine in the treatment of tics. Specific questions such as long term durability of beneficial effects, potential long-term side-effects, and comparisons to non-drug interventions are important, but not a focus of this pilot study.

The study will begin with a screening evaluation to ensure that each subject satisfies all eligibility criteria and to allow subjects to become familiar with our assessment procedures. Randomization of medications contained in look-alike capsules will occur at the baseline visit and is performed by a member of the Research Pharmacy staff. Patients will be evaluated at baseline, have direct formal scheduled evaluations at the end of treatment week's 2, 4, and 6 (+ 2 days), have telephone evaluations at the end of treatment week's 1, 3, and 5 (+ 2 days), and a final visit at 8 weeks. The primary outcome measure is effective tic suppression as determined by the difference in the Total Tic subscale (TTS) scores of the Yale Global Tic Severity Scale (YGTSS) at baseline and 6 weeks. Secondary outcome measures will include the change from baseline and 6 week scores for the YGTSS total score, the Clinical Global Impression -Improvement (CGI-I), and Patient Global Impression of Improvement (PGI-I). Secondary outcome for obsessive-compulsive behaviors will be measured by changes in the Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS). Safety measures will include the use of an expanded Pittsburgh Side Effect Scale modified to include side effects of riluzole and D-serine, incidence of adverse events, measurement of vital signs (BP, pulse) and body weight, physical examination, laboratory studies (comprehensive metabolic panel (CMP), complete blood count (CBC), plasma amino acids, and urine analysis), the DuPaul ADHD Rating Scale, Child Depression Inventory-short version (CDI-S), and Multi-Dimensional Anxiety Scale for Children (MASC). A Drug Safety Monitoring Board containing three clinician-scientists with experience in pharmacological trials will meet quarterly to review this study.

1. Study Population:

a) Recruitment: Subjects with TS/CMT (ages 8-17 years) will be recruited from the Tourette Syndrome Clinic at the Johns Hopkins Hospital and child psychiatry practice.

Patients with TS/CMT will be candidates for this study if: 1) they are tic-suppressing drug naive; 2) are not currently on treatment for TS (off medications for at least three weeks); or 3) if, in the judgment of the Investigators (Dr Singer and Grados), they are not adequately managed using current therapy (prescribed for greater than one month) and are willing to maintain a constant dose throughout the protocol. We believe that limiting the study to include only "drug-free" subjects would have a negative impact on recruitment. Many individuals with moderately severe to severe tics (TTS > 22) are receiving medications and in our opinion requiring prolonged tapers and extended drug free intervals are not in the best interest of the patient.

4. Procedures: i) Screening visit ( - 3 to -1 weeks): Determination of diagnostic eligibility criteria: medical history, complete physical examination (weight, heart rate, blood pressure, respiratory rate); familiarization with assessment procedures, rating scales for: tics, the Yale Global Tic Severity Scale (YGTSS), Clinical Global Impression-Severity Scale (CGI-S), obsessive-compulsive problems, Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS); attention deficit hyperactivity disorder, DuPaul ADHD Rating Scale, depression, Child Depression Inventory- Short Version (CDI-S); and anxiety, the Multidimensional Anxiety Scale for Children (MASC). Informed consent and child assent will be obtained. Urine (urine analysis) and blood (comprehensive metabolic panel, complete blood count, and plasma amino acids) will be obtained. Females who have begun to menstruate will be screened with a blood pregnancy test. Parents will be told the results of these tests. If the patient is uncomfortable with our telling the results of the pregnancy test to her parent(s), then they may decide not to take part in this study.

ii) Baseline Visit (Day 0): Determination of diagnostic eligibility criteria and the results of blood and urine analysis studies will be reviewed. Evaluation will include weight, heart rate, blood pressure, and respiratory rate, physical examination, rating scales for tics, obsessive-compulsive problems, ADHD, depression, and anxiety. As part of the baseline visit, the PI and Study Coordinator will meet with the parent to explain the procedures for dose titration, review in detail the outcome measures, and review approaches to administering medication (e.g., providing the pill with water or other beverage, observing the child swallow the medication without biting or chewing). Following confirmation of study eligibility, Dr Singer will forward a request for medication to the Johns Hopkins Research Pharmacy.

iii) Randomization (Day 0): A computer generated unequal randomized scheme will be used by a research pharmacist in the Johns Hopkins Research Pharmacy to assign patients to riluzole, D-serine, or placebo. The pharmacist making the treatment assignment will be proved with all essential data including patient name and study number, age, weight, and a list of concurrent medications. Subjects already on medications will be equally distributed among treatment groups. Twenty-four subjects each will be randomized to riluzole and D-serine and twelve to placebo. Medications, packaged in look-alike capsules, will be distributed by The Johns Hopkins Research Pharmacy. All medication codes will be retained by the research pharmacist until the completion of the study. All study medication will be double-blind: the Investigators, Study Coordinator and patient/parent will not be aware of the treatment assignment.

iv) Treatment groups (weeks 1 through 6): All treatments will be packaged in look-alike capsules. Patients will receive a 16 day supply of medication at the Baseline visit, and at the 2 and 4 week visits. Medications will be administered for the first week on a qday basis (morning) and thereafter on a twice a day schedule (morning and bedtime).

Each subject will be contacted at the end of weeks 1, 3, and 5 by telephone and evaluated in person end the end of weeks 2, 4, 6, and 8.

The maximum number of capsules per day in each treatment group is five. In order to achieve this fixed number, if necessary, Research Pharmacy will provide an additional vial of capsules containing the appropriate medication (see drug descriptions).

Riluzole (Rilutek):

Selection of dosage: For reference, in adults with ALS, riluzole was safe and effective in dosages of 100 and 200 mg twice daily. In a treatment study of infants with spinal muscular atrophy the maximum dosage was 10 mg higher than a 107 mg/m2 dose, e.g., for a 5 kg child whose surface area was 0.33 m2 , the dose was 35 mg/day. No child had any change in laboratory studies or had adverse effects.

Selection and timing of doses for subjects: The starting dose of riluzole will be 50 mg for one week; administered as one capsule (50) every morning. Dosage schedules will be flexible. If needed for tic suppression, the dose will be increased weekly by 50 mg and given in BID doses. The maximum dose will be 200 mg/day (administered as 2 capsules BID). In any individual subject, dose escalation may proceed more slowly, or the dose may be reduced if necessary. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing placebo (P) capsules. No changes in dosage will be made during the final week of treatment.

D-serine:

Selection of dosage: In man, D-serine is synthesized from L-serine via one enzymatic step catalyzed by the enzyme serine racemase. Levels of D-serine are controlled by the activity of serine racemase, the later having the highest expression in the forebrain. D-serine is currently being used in IND# 71,369 (D Javitt, PI). This approved serine will purchased by the Research Pharmacy at Johns Hopkins and encapsulated into capsules containing 250 and 500 mg of D-serine. The established treatment dose in the aforementioned IND is 30 mg/kg/day. In adults with schizophrenia and OCD, D-serine was safe and effective in dosages of 2 grams per day [Javitt Personal Communication].

Selection and timing of doses for subjects: The dosage schedule will be flexible with a maximum dose for each subject being 30 mg/kg/day. The following Table provides examples of subjects of different weights receiving increases of dosages. In any individual subject, dose escalation may proceed more slowly, or the dose may be reduced if necessary. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of capsules labeled as study drug, but containing either 250 (A) or 500 (B) mg tablets of D-serine or placebo (P); capsule content to be determined by patient's weight (see below). No changes in dosage will be made during the final week of treatment.

Placebo:

Placebo tablets will be formulated in look-alike capsules. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing additional placebo (P) capsules.

Compliance: To assess medication compliance, subjects and parents will be asked at each evaluation point (telephone and visit) about their compliance. Subjects will be required to return their medication vials at each visit and Dr Singer will verify whether the number of tablets returned by the subject corresponds to the prescribed intake. Compliance is defined as taking >80% to <120% of the prescribed doses.

vi) Concomitant medication: At each patient visit (baseline, 2, 4, and 6 weeks) the patient/parent will be asked to provide the names of any prescribed medications, over-the counter or herbal preparations used since the last visit.

vii) Medication taper: At the completion of the 6 week treatment phase, medication will be tapered over a ten day period; reduction of one capsule every other day. The half life of riluzole is 12 hours.

viii) Post-intervention (end of week 8) follow-up and management By the end of week 8, the subject will be completely off the study medication. Since study medications cannot be continued following completion of the protocol, this visit will, in part, be devoted to establishing ongoing care and treatment. All subjects will be offered ongoing care, treatment, and follow up with Dr Singer at Johns Hopkins. If the subject already has a treating physician, Dr Singer will be available to provide consultative services. Neither the Investigators nor subjects will receive information about the experimental drug assignment until the entire study has been completed.

ix) Evaluations: This is an 8-week study (6 weeks treatment, 2 week taper). Telephone evaluations will be performed by Dr Singer at the end of week's 1,3, and 5. At each telephone contact, clinical response, possible side effects, drug compliance, and medication adjustment will be discussed. Each subject will have direct evaluations by Dr Singer at baseline and the end of week's 2, 4, 6.and 8. These evaluations will include a pill count (except baseline) to assure compliance and safety measures including physical examination, vital signs (BP, heart rate), weight, blood and urine studies, and assessment of side effects using the Pittsburgh side effects scale. Dr Grados, a blinded outcome evaluator, will administer and score the outcome measures at each of the subject's visits (baseline, end of weeks 2, 4, 6).

x) Early stopping rules: Subjects may be withdrawn from the study at any time at the discretion of the subject, primary care physician, or Dr Singer.

1. Dr Singer can decide the subject should be withdrawn. This decision could be made because of an adverse effect, abnormal laboratory values, or a failure to comply with the study protocol.
2. The subject or his/her personal physician requests the subject be withdrawn.
3. The subject, for any reason, requires treatment with another therapeutic agent that could conflict with the use of riluzole or D-serine or complains of unacceptable side-effects.
4. A Drug Safety Monitoring Board (SMB). The duty of the SMB is to provide recommendations to the PI regarding medication issues and premature termination of the study for safety reasons. The SMB will be responsible for the quarterly review of data related to adverse clinical experiences and to assure that safety standards are maintained throughout the clinical trial. Three clinician-scientists, knowledgeable in the performance of clinical trials, members of the full time faculty at the adjacent Kennedy Krieger Institute, and not under the influence of the Johns Hopkins Director of Pediatric Neurology, will serve on the Board: Pediatric neurologists Dr's Gerald Raymond and Sakku Naidu and Dr Bruce Shapiro, a neurodevelopmental pediatrician.

The Research Coordinator, with assistance of the Statistician, will prepare data for the quarterly review by the SMB from data stored on a secure computer. The SMB will act independently to review the data. If there is any safety concern related to one or more of these groups, then the Board may choose to identify the actual treatment groups by access to the randomization codes maintained by the pharmacy. Significant adverse events will be reported to the IRB, SMB and FDA within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Tourette syndrome (criteria based on the TS Classification Study Group), which includes onset before 18 years, multiple involuntary motor tics, one or more vocal tics, a waxing and waning course, the gradual replacement of old symptoms with new ones, the presence of tics for more than one year, the absence of other medical explanations (effects of a substance (e.g., stimulants) or a general medical condition for tics, and observation of tics by a reliable examiner) or Chronic Motor Tic disorder (criteria similar to Tourette syndrome except for the absence of vocal tics)
* Age 8-17 years, either gender
* Observable tics, achieving a minimum score of > 22 on the Total Tic score of Yale Global Tic Severity Scale (YGTSS)
* Tic symptoms severe enough to warrant therapy (e.g., causing psycho-social or physical difficulty)
* Written informed consent provided by the patient's parent (or legal guardian) and assent provided by the patient consistent with Institutional Review Board requirements
* Ability and willingness to comply with study protocol requirements
* Women of childbearing potential must be using a medically acceptable contraceptive method. Acceptable methods of birth control are limited to: Intra-Uterine Device (IUD), oral, implantable, injectable contraceptives and estrogen patch, double barrier method (spermicide+diaphragm), or abstinence
* Baseline weight of at least 33 kilograms
* Tic-suppressing drug naive, or currently not on treatment for TS (off medications for at least three weeks), or if, in the judgment of the PI, they are not adequately managed using current therapy (prescribed for greater than one month) and are willing to maintain a constant dose throughout the protocol.

Exclusion Criteria:

* Secondary tics
* Significant medical illness (metabolic, endocrine, cardiac, hematological, gastrointestinal, pulmonary, epilepsy)
* Current major depression
* generalized anxiety disorder
* separation anxiety disorder
* psychotic symptoms (based on clinical evaluation and the results of the CY-BOCS, CDI-S, and MASC evaluations)
* pervasive developmental disorder
* autism
* mental retardation (I.Q. less than 70)
* anorexia/bulimia, or substance abuse
* Any other conditions that in the opinion of the Investigators would interfere with the evaluation of the results or constitute a health hazard for the patient
* Pregnancy
* Hypersensitivity to D-serine or riluzole
* Abnormal laboratory values on screening laboratory testing if clinically significant at the Principal Investigator's discretion.

Subjects with co-morbid ADHD, obsessive compulsive disorder (OCD), and conduct disorder will not be excluded as long as these diagnoses are not the subject's primary problem

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey S Singer, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consent will be obtained by Dr. Harvey Singer from eligible patients at the Tourette Syndrome Clinic in the JHH Outpatient Center. Patients will be given a general synopsis of the research study and carefully explained each page of the consent form. Once informed consent is obtained, the subject will be considered to have entered the study.
Pre-assignment Details: 39 patients were enrolled at a screening visit, but for a variety of reasons (i.e. no longer interested, concerned about blood draws, medication use, et cetera) only 30 started medications at the baseline visit. Of these 30, 24 completed the study.
Period: Overall Study
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Started | 12 | 12 | 6
Completed | 9 | 10 | 5
Not Completed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo | Total
Number analyzed (Participants) | 9 | 10 | 5 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (3.04) | 13.1 (1.98) | 12.6 (2.76) | 13.5 (2.58)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 10 | 5 | 24
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 0 | 3
  Male | 6 | 10 | 5 | 21
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to 6-week Scores for The Total Tic Subscale (TTS)
Description: The primary outcome measure is effective tic suppression as determined by the difference in the Total Tic subscale (TTS) scores of the Yale Global Tic Severity Scale (YGTSS) at baseline and 6 weeks.
  i) Yale Global Tic Severity Scale (YGTSS): The YGTSS is a semi-structured clinical interview designed to measure current tic severity. It is comprised of two parts, a tic score (0-50) and a total impairment score (0-50). The Total Tic Score (TTS: 0-50) has been selected as the primary outcome measure. The scale ranges from 0 (the best possible outcome) to 50 (the worst possible outcome). This scale is considered the best currently available scale to rate the severity of tics. The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6.
Time Frame: Baseline and 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 6.2 (8.1) | 10.5 (7.2) | 10.2 (4.3)

2. Secondary Outcome: The Change From Baseline to 6-week Scores for the Yale Global Tic Severity Scale (YGTSS) Total Score.
Description: i) Yale Global Tic Severity Scale (YGTSS): The YGTSS is a semi-structured clinical interview designed to measure current tic severity. It is comprised of two parts, a tic score (0-50) and a total impairment score (0-50), total maximum score is 100. This scale has established validity, as assessed by Dr. Walkup and colleagues and is considered the best currently available scale to rate the severity of tics. This scale ranges from 0 (the best possible outcome) to 100 (the worst possible outcome).
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6. Please note that summary data (mean and standard deviation per group) were intended to be reported, and not participant level data (i.e. each individual data point of every subject per group).
Time Frame: Baseline and 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 22 (16.3) | 23.5 (11.5) | 19.4 (10.6)

3. Secondary Outcome: The Change From Baseline to 6-week Score for the Clinical Global Impression -Improvement (CGI-I).
Description: Clinical Global Impression-Improvement (CGI-I): The CGI-I is used to compare current severity to baseline. A score of 1 corresponds to "very much improved"; 2 equals "much improved;" 3 denotes "minimal change"; and 4 represents "no change." Scores above 4 are used to indicate deterioration, i.e., 5 equals "minimally worse;" 6 is "much worse;" and 7 is "very much worse."
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6. Please note that summary data (mean and standard deviation per group) were intended to be reported, and not participant level data (i.e. each individual data point of every subject per group).
Time Frame: Baseline and 6-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 0.78 (0.83) | 1.70 (0.67) | 1 (1)

4. Secondary Outcome: The Change From Baseline to 6-week Score for the Patient Global Impression of Improvement (PGI-I).
Description: Patient Global Impression of Improvement (PGI-I) is a single seven point scale in which the patient/parent is asked to assess the change in overall condition ranging from "very much" improved to "very much worse."
  A score of 1 corresponds to "very much better"; 2 equals "much better;" 3 denotes "a little better"; and 4 represents "no change." Scores above 4 are used to indicate deterioration, i.e., 5 equals "a little worse;" 6 is "much worse;" and 7 is "very much worse."
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6. Please note that only summary data (mean and standard deviation per group) were intended to be reported, and not participant level data (i.e. each individual data point of every subject per group)--this applies to all outcome measures reported in the results.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | -0.56 (0.88) | -0.10 (0.88) | 0.60 (1.14)

5. Secondary Outcome: Changes in the Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) From Baseline to 6-weeks.
Description: Secondary outcome for obsessive-compulsive behaviors will be measured by changes in the Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) from baseline to 6-weeks.
  The severity of OCD was evaluated using either the Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS) or Yale-Brown Obsessive Compulsive Scale (Y-BOCS). The (C)Y-BOCS is the most widely used instrument to assess the severity of obsessive-compulsive symptoms in research studies involving children. The (C)Y-BOCS has well established psychometric properties. The scale ranges from 0 (the best possible outcome) to 10 (the worst possible outcome).
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6.
Time Frame: Baseline and 6-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 5.9 (6.0) | 1.8 (5.8) | -0.8 (4.0)

6. Secondary Outcome: The Change From Baseline to 6-week in Plasma Amino Acid Levels
Description: Blood testing was performed at baseline and at each clinic visit. Data shown below reflects baseline Glutamic Acid minus Week 6 Glutamic Acid, and baseline Serine minus Week 6 Serine levels; as acquired from the blood tests during these respective clinic visits.
Time Frame: Baseline and 6 weeks.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
micromol/L
  Baseline Glutamic Acid Minus Week6 Glutamic Acid | 1.56 (30.55) | 23.20 (39.07) | 10.20 (22.88)
  Baseline Serine Minus Week6 Serine | -108.22 (69.38) | 13.30 (30.29) | -4.40 (25.21)

7. Secondary Outcome: The Change From Baseline to 6-week in Scores of the DuPaul Attention Deficit Hyperactivity Disorder Rating Scale.
Description: DuPaul ADHD Rating Scale: The presence of ADHD symptoms will be assessed using the DSM-IV version of the ADHD rating scale developed by DuPaul. This scale has been normed in large clinical and community samples and has excellent psychometric properties including a test-retest reliability over a 2-week period of 0.93 and significant correlations with direct observations of classroom behavior. The scale has a maximum possible score of 72, and a minimum of 0. The scale ranges from 0 (the best possible outcome) to 70 (the worst possible outcome).
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6.
Time Frame: Baseline and 6 weeks
Population: Please note that one subject failed to complete this assessment on week 6; therefore, the total number of participants in the placebo group for DuPaul ADHD is 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 12 subjects age 8-17 years with moderate to severe TS (TTS > 22) will be enrolled in this treatment arm. They will receive placebo for 6-weeks of the study, during which time drug dose may gradually be increased as needed. At 6-weeks participants will taper off drug.
  Placebo: Placebo tablets will be formulated in look-alike capsules. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing additional placebo capsules.
  Please note that one subject failed to complete this assessment on week 6; therefore, the total number of participants in the placebo group for DuPaul ADHD is 4.
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 4
units on a scale | 4.56 (12.17) | 5.10 (10.05) | -7.00 (4.39)

8. Secondary Outcome: The Change From Baseline to 6-week in Scores of the Child Depression Inventory - Short Version (CDI-S) Scale
Description: Depression Inventory-Short Version (DI-S): Depression severity will be rated by using the Depression Inventory-Short Version (DI-S). This 10 item scale takes about 5 minutes to complete. It has excellent psychometric properties and is designed for repeated administrations over time. The maximum possible score of 20, and a minimum score of 0. Higher score on this scale indicates greater severity of depression in children.
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 3). For consistency, all values weather positive or negative represent baseline minus week 6.
Time Frame: Baseline and 6-weeks
Population: Please note that two subjects failed to complete this assessment on week 6; therefore, the total number of participants in the placebo group for CDI-S is 3.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: 12 subjects age 8-17 years with moderate to severe TS (TTS > 22) will be enrolled in this treatment arm. They will receive placebo for 6-weeks of the study, during which time drug dose may gradually be increased as needed. At 6-weeks participants will taper off drug.
  Placebo: Placebo tablets will be formulated in look-alike capsules. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing additional placebo capsules.
  Please note that two subjects failed to complete this assessment on week 6; therefore, the total number of participants in the placebo group for CDI-S is 3.
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 3
units on a scale | 0 (3.0) | -0.1 (0.9) | 1.0 (2.6)

9. Secondary Outcome: The Change From Baseline to 6-week in Scores of the Multi-Dimensional Anxiety Scale for Children (MASC)
Description: Multidimensional Anxiety Scale (MAS): Anxiety will be followed using the Multidimensional Anxiety Scale for Children (MASC), which has been developed by Dr. John March at Duke University and is now considered the preferred instrument for rating anxiety. The MASC asks the patient how they have been thinking and acting recently. It has a maximum possible score of 117 and a minimum score of 0. Higher score on this scale indicates greater severity of anxiety in children.
  The data provided below represents the mean change (baseline minus six week) for the D-serine group (n = 9), Riluzole (n = 10), and Placebo group (n = 5). For consistency, all values weather positive or negative represent baseline minus week 6.
Time Frame: Baseline and 6-weeks
Population: Please note that one subject failed to complete this assessment on week 6; therefore, the total number of participants in the placebo group for MASC is 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 12 subjects age 8-17 years with moderate to severe TS (TTS > 22) will be enrolled in this treatment arm. They will receive placebo for 6-weeks of the study, during which time drug dose may gradually be increased as needed. At 6-weeks participants will taper off drug.
  Placebo: Placebo tablets will be formulated in look-alike capsules. At the 4 week visit, if an additional dosage increase is prescribed by Dr Singer, the pharmacy will provide an additional vial of 14 capsules labeled as study drug, but containing additional placebo capsules.
  Please note that one subject failed to complete this assessment on week 6; therefore, the total number of participants in the placebo group for MASC is 4.
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 4
units on a scale | 1.33 (14.44) | -3.30 (6.98) | 6.25 (6.28)

10. Secondary Outcome: Expanded Pittsburgh Side Effect Scale Modified to Include Side Effects of Riluzole and D-serine.
Description: The scale consists of 25 items with a score of 0 to 3 per item. 0- none, 1- mild, 2- moderate and 3- severe side effect. The total could be zero (no side effects) to 75 or higher.The scale also allows for the addition of other side effects not included in the original scale and the total score could potentially be higher than 75. If no other side effects outside of the original scale are recorded, the the maximum score remains at 75.
Time Frame: Baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 0.56 [0 to 75] | 0.5 [0 to 75] | 0.2 [0 to 75]

11. Secondary Outcome: Expanded Pittsburgh Side Effect Scale Modified to Include Side Effects of Riluzole and D-serine.
Description: as for outcome 10
Time Frame: Week 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 0.33 [0 to 75] | 0 [0 to 75] | 0 [0 to 75]

12. Secondary Outcome: Expanded Pittsburgh Side Effect Scale Modified to Include Side Effects of Riluzole and D-serine.
Description: as for outcome 10
Time Frame: Week 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 0.22 [0 to 75] | 0.5 [0 to 75] | 0.25 [0 to 75]

13. Secondary Outcome: Expanded Pittsburgh Side Effect Scale Modified to Include Side Effects of Riluzole and D-serine.
Description: as for outcome 10
Time Frame: Week 6
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 0.44 [0 to 75] | 0.5 [0 to 75] | 0.5 [0 to 75]

14. Secondary Outcome: Expanded Pittsburgh Side Effect Scale Modified to Include Side Effects of Riluzole and D-serine.
Description: as for outcome 10
Time Frame: Week 8
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Number analyzed (Participants) | 9 | 10 | 5
units on a scale | 0.33 [0 to 75] | 0.2 [0 to 75] | 0.2 [0 to 75]

ADVERSE EVENTS:
Arm/Group | D-serine (Glutamate Agonist) | Riluzole (Glutamate Antagonist) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/5

LIMITATIONS AND CAVEATS:
Study was limited by its small sample size as well as a small placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No